CLINICAL TRIAL: NCT00846339
Title: [11C] Raclopride PET Imaging Study That Investigates Relation Between Occupancy of Dopamine D2 Receptors and Genotypes of DRD2 After Bupropion Administration
Brief Title: PET Imaging Study on Occupancy of Dopamine D2 Receptors and Genotypes After Bupropion Administration
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Ministry of Health, Welfare and Family Affairs (Unknown); Korea National Enterprise for Clinical Trials (Other)
Responsible Party: Kyung-Sang Yu, Seoul National University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SNUCPT08_BUP1
Record Dates: First submitted 2009-02-14; First posted 2009-02-18 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2011-02

CONDITIONS: Smoking
Keywords: Smoking cessation; Bupropion
MeSH Terms: conditions — Smoking; Smoking Cessation | interventions — Bupropion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): DRD2 Taq1A1 allele
  Interventions: Drug: Bupropion
- 2 (Experimental): DRD Taq1 A2 homozygote2
  Interventions: Drug: Bupropion

INTERVENTIONS:
Drug: Bupropion — bupropion

SUMMARY:
Bupropion has different effects on D2 dopamine receptors according to genotype.

DETAILED DESCRIPTION:
Open, one arm, single sequence, 2-period, study stratified into 2 DRD2 genotype groups For subjects who volunteer to cease smoking, genotypes are investigated. Twelve subjects are enrolled (6 - DRD2 Taq1A1 allele, 6 - DRD2 Taq1A2 homozygotes). Subjects receive baseline raclopride PET (High Specific Activity, Low Specific Activity).

* Period 1 Subjects receive 150 mg of bupropion SR every day. After 1 week of medication, pharmacokinetic and PET studies are performed.
* Period 2 Subjects receive 150 mg of bupropion SR twice a day. After 1 week of medication, pharmacokinetic and PET studies are performed.

ELIGIBILITY:
Inclusion Criteria:

* Active smoker (more than 10 cigarettes per day for the past 2 years)

Exclusion Criteria:

* Medical or psychiatric co-morbidity
* Hypersensitive to bupropion

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2008-11; Primary Completion 2009-03 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Dopamine receptor occupancy | 1 week

SECONDARY OUTCOMES:
Pharmacokinetic parameters of bupropion and hydroxybupropion | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Sang Yu, MD, Principal Investigator — Seoul National Univeristy Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea